CLINICAL TRIAL: NCT06935071
Title: Endoprosthetic Replacement for Pathological Fractures of the Hip: A 35-year Update
Status: Active, not recruiting | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 16-1122
Record Dates: First submitted 2025-04-11; First posted 2025-04-18 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Hip Fractures; Hip Fracture Pathologic; Pathological Fracture; Pathological Fracture of Hip
Keywords: hip fractures; pathological hip fractures; hip fracture parthologic; pathological fracture of hip; 16-1122; Memorial Sloan Kettering Cancer Center
MeSH Terms: conditions — Hip Fractures; Fractures, Spontaneous | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants who received endoprosthetic reconstruction: Participants have received endoprosthetic reconstruction for pathologic fracture of the proximal femur.
  Interventions: Other: Data Collection and Analysis

INTERVENTIONS:
Other: Data Collection and Analysis — Patient data will be analyzed to ensure that all data fields are available and that suitable sample size is available to answer the research objectives. The rate of ambulation at discharge, ambulation at 3 month follow up (if available), time to death, and pain score between the historic cohort with a current cohort of patients will be compared.

SUMMARY:
This study will be based on a retrospective review of patients who received endoprosthetic reconstruction for pathologic fracture of the proximal femur. The objectives would be two-fold: (1) to compare rates ofambulation, pain, and survival to the historic cohort and (2) to identify predictors of ambulation in the current population.

ELIGIBILITY:
Inclusion Criteria:

* Participants have received endoprosthetic reconstruction for pathologic fracture of the proximal femur

Exclusion Criteria:

* Participants with fractures greater than 3mm from the lesser trochanter
* Participants without histopathologic confirmation of tumor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: For this retrospective data review, the study team will query the orthopaedic caisis database and IDB to obtain a list of all participants who have received endoprosthetic reconstruction for pathologic fracture of the proximal femur.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2016-08-04 (Actual); Primary Completion 2026-08-04 (Estimated); Study Completion 2026-08-04 (Estimated)

PRIMARY OUTCOMES:
Comparison of rates of ambulation, pain, and survival to the historic cohort | up to 10 years
  This study will be based on a retrospective review of patients who received endoprosthetic reconstruction for pathologic fracture of the proximal femur.

CONTACTS AND LOCATIONS:
Overall Officials: John Healey, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
• Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org